CLINICAL TRIAL: NCT05953298
Title: Evaluation by Electrical Impedancemetry of the Variation of Lung Volumes Under NIV in Patients With COPD
Brief Title: Evaluation by Electrical Impedancemetry of the Variation in Lung Volumes Under Non-invasive Ventilation (NIV) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: Eval 3V-BPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2023/10
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease; non invasive ventilation; end-expiratory lung volume; electrical impedance tomography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with COPD (Experimental): Patients with COPD in stable condition fitted with long-term NIV
  Interventions: Device: Electrical impedance tomography (EIT)

INTERVENTIONS:
Device: Electrical impedance tomography (EIT) — Electrical impedance tomography (EIT) is a non-invasive evaluation tool, without radiation, simple to set up at the patient's bedside and validated, making it possible to monitor the distribution of ventilation and lung recruitment with high temporal resolution, dynamic way and at a regional level

SUMMARY:
The aim of this physiologic research is to assess lung volumes variations under NIV in stable COPD patients to understand the impact of "high-intensity" ventilation following the current recommendations. The main objective is to evaluate the variation of End-expiratory lung volume (EELV) reflecting the functional residual capacity (FRC), via the End-tidal lung impedance (EELI) obtained by electrical impedance tomography during a 20 minutes NIV session.

DETAILED DESCRIPTION:
In patients with COPD, European recommendations recommend the use of NIV with a "high pressure" setting (1). These ventilatory modalities go against what is done in acute. Indeed, in this case, the pressures are much lower, because the risk of asynchronies and dynamic hyperinflation under NIV is then very important.

The usual techniques for evaluating lung volume and dynamic hyperinflation do not allow this to be measured under NIV.

Assessing lung volumes under NIV in stable COPD patients is therefore of major interest in understanding the impact of "high-intensity" ventilation.

Electrical impedance tomography (EIT) is a non-invasive evaluation tool, without radiation, simple to set up at the patient's bedside and validated, making it possible to monitor the distribution of ventilation and lung recruitment with high temporal resolution, dynamic way and at a regional level.(2) Among these measures, the End-Expiratory Lung Impedance (EELI), strongly correlated to the End-Expiratory Lung Volume (EELV), is the reflection of the FRC and can be dynamically monitored in real time at the patient's bedside(3). However, it has never been used in stable COPD patients on NIV, and could be an interesting tool for analyzing the impact of NIV on lung volumes.

The main objective is to evaluate the variation of EELV reflecting the functional residual capacity (FRC), via the End-tidal lung impedance (EELI) obtained by electrical impedance tomography, during a 20-minute session of NIV in patients with COPD at the stable state

The secondary objectives will be:

* To evaluate the variation of the EELV reflecting the FRC, via the EELI obtained by electrical impedance tomography, before, during and after a 20-minute session of NIV in stable-state COPD patients.
* Evaluate the relationship between the variation of PtCO2, and that of EELV under NIV, reflection of the FRC, via the EELI obtained by electrical impedance tomography.
* Identify responder and non-responder patient subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD in stable condition fitted with long-term NIV followed at Bordeaux University Hospital;
* Patient benefiting from social protection from the national health insurance fund;
* Patient having read the patient information letter and given his non-objection to participate in the study.

Exclusion Criteria:

* Obesity with a BMI > 35;
* Respiratory exacerbation during treatment;
* Patient with one or more contraindications to the implementation of EIT(7):

  * Pacemaker, defibrillator, electric active medical device;
  * Damaged skin condition, dressing on the observation area;
  * Risk related to fitting the belt (fracture, spinal lesions, etc.);
  * Uncontrollable movements;
  * Current electrotherapy;
  * Presence of a magnetic field (magnetic resonance imaging);
  * Other bioimpedance measurements in progress;
  * Pregnant woman ;
  * Tidal volume < 1ml/kg;
* Patient having read the patient information letter and refusing to participate in the study (Loi Jardé research category 3);
* Patient under guardianship, curatorship, or deprived of freedom of administrative or judicial decision;
* Patient included in other protocols that may interact with this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
End-Expiratory Lung Impedance (EELI) evolution during NIV sessions | Day 1
  End-Expiratory Lung impedance is related to the End-Expiratory Lung Volume reflecting the functional residual capacity (FRC). It is obtained by electrical impedance tomography. EELI values are presented in arbitrary values (v.a) and can vary greatly between individuals. Thus, as previously proposed by (4), the EELI values during the different measurement phases will be assessed and presented as a percentage change from their reference value. The main objective of this study aims to observe the evolution of the EELI under NIV in stable COPD patients, the reference EELI value will be that measured at T1 (NIV initiation+1 minute), compared to that measured at T2 (NIV+20minutes) under the ∆EELI%T2 abbreviation from the following calculation: ∆EELI%T2 = (EELIT1-EELIT2)/EELIT1*100

SECONDARY OUTCOMES:
End-Expiratory Lung Impedance (EELI) evolution before, during and NIV sessions | Day 1
  A secondary objective of this research is to observe the evolution of the EELI before, during and after the NIV. In this context, the reference value will be the measurement of the EELI before the NIV, i.e. EELIT0. Thus the EELI values at T1 (NIV initiation+1 minute), T2 (NIV+20minutes) and T3 (5minutes after NIV) will be presented as a percentage change compared to T0 and will be respectively ∆EELI%T1, ∆EELI %T2 and ∆EELI%T3, respecting the following calculation: ∆EELI%Tx = (EELIT0-EELITx)/EELIT0*100.
Transcutaneous capnia | Day 1
  A secondary objective of this research is to observe the evolution of transcutaneous capnia (PtCO2) in mmHg via a capnograph before (T0), during (T1, T2) and after NIV (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Leo GRASSION, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Haut Lévêque, Centre Hospitalier Universitaire de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarz SB, Magnet FS, Windisch W. Why High-Intensity NPPV is Favourable to Low-Intensity NPPV: Clinical and Physiological Reasons. COPD. 2017 Aug;14(4):389-395. doi: 10.1080/15412555.2017.1318843. Epub 2017 May 11. PMID 28494170
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Hinz J, Hahn G, Neumann P, Sydow M, Mohrenweiser P, Hellige G, Burchardi H. End-expiratory lung impedance change enables bedside monitoring of end-expiratory lung volume change. Intensive Care Med. 2003 Jan;29(1):37-43. doi: 10.1007/s00134-002-1555-4. Epub 2002 Nov 20. PMID 12528020
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805